CLINICAL TRIAL: NCT02218034
Title: Safety, Tolerability and Pharmacokinetics of AGN-190168 in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 190168-069
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AGN-190168 Formulation 1 (Experimental): AGN-190168 Formulation 1 applied topically to the face, neck, upper chest, upper back, and shoulders once daily for 29 days.
  Interventions: Drug: AGN-190168 Formulation 1
- AGN-190168 Formulation 2 (Experimental): AGN-190168 Formulation 2 applied topically to the face, neck, upper chest, upper back, and shoulders once daily for 29 days.
  Interventions: Drug: AGN-190168 Formulation 2
- TAZORAC® Gel 0.1% (Active Comparator): TAZORAC® Gel 0.1% (tazarotene gel 0.1%) applied topically to the face, neck, upper chest, upper back, and shoulders once daily for 29 days.
  Interventions: Drug: tazarotene gel 0.1%
- TAZORAC® Cream 0.1% (Active Comparator): TAZORAC® Cream 0.1% (tazarotene cream 0.1%) applied topically to the face, neck, upper chest, upper back, and shoulders once daily for 29 days.
  Interventions: Drug: tazarotene cream 0.1%

INTERVENTIONS:
Drug: AGN-190168 Formulation 1 — AGN-190168 Formulation 1 applied topically to the face, neck, upper chest, upper back, and shoulders once daily for 29 days.
  Arms: AGN-190168 Formulation 1
Drug: AGN-190168 Formulation 2 — AGN-190168 Formulation 2 applied topically to the face, neck, upper chest, upper back, and shoulders once daily for 29 days.
  Arms: AGN-190168 Formulation 2
Drug: tazarotene gel 0.1% — Tazarotene gel 0.1% applied topically to the face, neck, upper chest, upper back, and shoulders once daily for 29 days.
  Other Names: TAZORAC® Gel 0.1%
  Arms: TAZORAC® Gel 0.1%
Drug: tazarotene cream 0.1% — Tazarotene cream 0.1% cream applied topically to the face, neck, upper chest, upper back, and shoulders once daily for 29 days.
  Other Names: TAZORAC® Cream 0.1%
  Arms: TAZORAC® Cream 0.1%

SUMMARY:
This is a safety, tolerability and pharmacokinetics study of AGN-190168 in subjects with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acne vulgaris on the face
* No tobacco use for the past 30 days, and willing to refrain from nicotine use during the study
* Willing to avoid excessive or prolonged exposure of the treated skin to ultraviolet light (eg, sunlight, tanning beds) and extremes in weather, such as wind or cold, throughout the study
* If male, willing to maintain routine shaving regimen for the duration of the study and avoid shaving 12 hours prior to specified visits
* Females of childbearing potential must use a reliable method of contraception

Exclusion Criteria:

* Use of phototherapy devices (eg, ClearLight™) and adhesive cleansing strips (eg, Ponds® and Biore®), as well as cosmetic procedures (eg, facials, peeling, and comedone extraction) in the area to be treated in the past 1 week
* Use of topical anti-inflammatory drugs, salicylic acid (eg, Clearasil® and Clean & Clear®), corticosteroids, antibiotics, antibacterials (including benzoyl peroxide-containing products [eg, benzamycin]), retinoids, and other topical acne treatments (eg, photodynamic therapy, laser therapy, and medicated soaps) in the area to be treated in the past 2 weeks
* Ability to abstain from caffeine-containing products on the dates instructed

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Level (Cmax) of AGN-190168 | Day 29
Maximum Plasma Level (Cmax) of AGN-190168 Metabolite | Day 29
Local Dermal Tolerability as Assessed by the Subject Using a 4-Point Scale | Day 29
Local Dermal Tolerability as Assessed by the Investigator Using a 4-Point Scale | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- College Station, Texas, United States